CLINICAL TRIAL: NCT05156242
Title: Corticospinal and Motor Behavior Responses After 6-week Transcranial Direct Current Stimulation and Neuromuscular Electrical Stimulation Combined With Motor Control Exercises in Patients With Chronic Low Back Pain
Brief Title: Corticospinal and Motor Behavior Responses After Physical Therapy Intervention in Patients With Chronic Low Back Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: University of South Carolina (Other)
Responsible Party: Principal Investigator, Peemongkon Wattananon, Assistant Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MU-CIRB 2021/327.2906
Record Dates: First submitted 2021-12-01; First posted 2021-12-14 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Low Back Pain
Keywords: Low back pain; Corticospinal excitability; Transcranial magnetic stimulation; Transcranial direct current stimulation; Neuromuscular electrical stimulation; Motor control exercise; Lumbar multifidus muscle
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: 4-arm randomized controlled trial (active-tDCS priming MCE, sham-tDCS priming MCE, NMES priming MCE, and conventional physical therapy)
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participant will be blinded using active vs sham intervention. Care provider is not involving in data collection and blinded to type of stimulation.
  Outcomes assessor will be blinded to the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Active-tDCS priming MCE (Experimental): The subjects in active-tDCS priming with MCE group will receive the tDCS using 5X7 cm electrodes in which anodal electrode will be placed on M1 representing the back muscles (1 cm anterior and 4 cm lateral to the vertex), while cathodal electrode will be placed on contralateral supraorbital area. The intensity will be set at 2 mA with 10-second fade in/out. The subject will be stimulated by tDCS for 20 minutes. After that, the subjects will receive 20-minute MCE.
  Interventions: Device: Active-tDCS priming MCE
- Sham-tDCCS priming MCE (Sham Comparator): The subjects in sham-tDCS priming with MCE group will receive a 20-minute sham tDCS by setting the intensity at zero mA. After that, the subjects will receive 20-minute MCE.
  Interventions: Device: Sham-tDCS priming MCE
- NMES priming MCE (Active Comparator): The subjects in NMES priming with MCE group will receive the NMES using interferential mode (6000 Hz, beat frequency 20-50 Hz, scanning effect) on bilateral LM. The intensity will be set at the subject's maximum tolerance. Stimulation will be set at 10 seconds on and 60 seconds off to minimize muscle fatigue. The total NMES time is 20 minutes. After that, the subjects will receive 20-minute MCE.
  Interventions: Device: NMES priming MCE
- Conventional physical therapy (Active Comparator): The subjects in conventional physical therapy group will receive physical therapy modality (e.g., ultrasound, TENS, etc.) and general exercises.
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Device: Active-tDCS priming MCE — tDCS is used to enhance cortical excitability before motor control exercises.
  Other Names: MINDD STIM, Ybrain Inc., Korea
  Arms: Active-tDCS priming MCE
Device: Sham-tDCS priming MCE — tDCS will be set at 0 mA for 20 minutes before motor control exercise.
  Other Names: MINDD STIM, Ybrain Inc., Korea
  Arms: Sham-tDCCS priming MCE
Device: NMES priming MCE — NMES is used to enhance lumbar multifidus motor unit recruitment before motor control exercise.
  Other Names: Sonopuls-490 combination therapy, Enraf-Nonius BV, The Netherlands
  Arms: NMES priming MCE
Other: Conventional physical therapy — Conventional physical therapy includes modality for pain control, general exercise to improve muscle strength, endurance, and flexibility, and functional training (sit to stand, walking, etc.).
  Arms: Conventional physical therapy

SUMMARY:
This study aims to 1) determine the immediate effects of transcranial direct current stimulation (tDCS) on corticospinal excitability, lumbar multifidus muscle (LM) activation, as well as lumbar stability in patients with chronic low back pain (CLBP), 2) determine the immediate effects of neuromuscular electrical stimulation (NMES) on corticospinal excitability, LM activation, as well as lumbar stability in patients with CLBP, 3) compare the effectiveness of 6-week intervention program among tDCS priming with motor control exercise (MCE), NMES priming with MCE, and MCE alone in patients with CLBP, and 4) determine the associations among corticospinal excitability, LM activation, lumbar stability, movement patterns, and clinical outcomes in patients with CLBP.

DETAILED DESCRIPTION:
This proposed study will use a sample of convenience between the ages of 18 and 40. Subjects who has low back pain more than 3 months or a recurrent pattern of low back pain at least two episodes that interfered with activities of daily living and/or required treatment will be recruited by flyers posted in 2 university physical therapy clinics, as well as word of mouth from subjects and friends. Subjects without a history of low back pain in lifetime will be also recruited to establish normative data. Subjects who are interested in participation will undergo a screening process using inclusion-exclusion criteria checklist and receive brief information regarding the study. If they meet all inclusion criteria, the consent process will be performed.

All subjects will fill out the information sheet for demographic data. Subjects in CLBP will undergo standardized movement system impairment examination and transverse abdominis muscle thickness measurement, self-report questionnaires; pain, disability, quality of life, and fear of movement) and functional tests (5-time sit to stand test, 2-minute step test, functional reach test, prone trunk extension test and abdominal curl test). The project manager responsible for organizing the data collection and blindness will arrange the appointments with the subjects for 2 biomechanical data collection. For the subjects who refuse to participate in biomechanical lab testing, they will proceed to 6-week intervention.

In the first visit (pre-intervention visit#1), biomechanical data including motion and clinical data, lumbar stability, and cortical excitability will be collected. The body landmarks will be identified. These landmarks include 1) lumbar spinous process of T12-S2, 2) lumbar erector spinae (ES) and multifidus (LM) (3 cm lateral to L3 spinous process and 2 cm lateral to L3 spinous process, respectively), 3) bilateral lateral epicondyle of femur, and 4) bilateral lateral malleolus. Spinous process of L1, S2, bilateral lateral epicondyle of femur, and bilateral lateral malleolus will be used as locations for motion tracking sensors, while ES and LM location will be used to place surface electrode for cortical excitability measurement.

For motion and clinical observation data collection, subjects will be instructed to perform 1) sustained positions including usual sitting, corrected position in sitting, usual standing, corrected position in standing, as well as 2) functional movements including active forward bend, stand to sit, sit to stand, walking for 30 seconds, stair ascending, stair descending, and pick up a box from the floor. Then, the subjects will be asked to perform clinical movement tests including active forward bend (waiter's bow), standing with posterior tilt, single leg stance on left and right foot, single leg squat on left and right leg, supine with right and left straight leg raise tests, supine with right and left hip abduction with knee flexion tests, quadruped backward rock test, prone with right and left knee flexion tests, prone with right and left hip internal/external rotation tests, prone with right and left hip extension tests. 1-2 repetitions of practice trial will be provided to familiarize with the movement. Each subject performs 2 sets of 3 consecutive repetitions of each functional movement and clinical movement test in fixed order, while 2 assessors independently rate presence/absence of aberrant movement. Thirty-second rest will be provided between movement tests (rest period can be longer if necessary). Pain intensity, heart rate and rating of perceive exertion (RPE) will be monitored after each test. Motion sensors will be removed.

After that, subjects will undergo lumbar stability test. Two electromagnetic tracking sensors will be placed on T12 and S2 spinous processes, while one sensor will be attached to hand-held dynamometer. Subjects will be asked to position in prone on the treatment bed with both feet on the floor. A researcher will apply 10-kg compression force on L1 to L5 spinous processes for 2 seconds. This 10-kg compression force is derived from the pilot work in which the researchers plotted the graph between compression force in X-axis and posteroanterior displacement in Y-axis. The graph demonstrated plateau (no displacement even increasing in compression force) at approximately 10 kg. Then, subjects will be asked to lift both legs away from the floor presumably activating LM, while the researcher re-apply the same compression force on L1 to L5 again. Pain will be recorded when applying compression force on each spinal level. Sensor displacement will be collected to represent lumbar stability.

For cortical excitability measurement, the subjects will undergo corticospinal excitability measurement using transcranial magnetic stimulation (TMS). The researcher will use ES and LM landmarks for EMG electrode placement. Before placing surface EMG electrodes, the skin will be lightly abraded using abrasive paper and cleaned using cotton with alcohol to lower the skin impedance. Electrodes will be aligned parallel to the muscle fibers. Then, Subjects seat comfortably in a reclined chair with both arms supported. They will be asked to wear a swim cap used to identify stimulation areas for ES and LM. The researcher uses TMS with single-pulse monophasic to stimulate each point over pre-marked scalp sites on a 5 X 7 grid (0-5 cm lateral and from 5 cm anterior to 2 cm posterior to the vertex). Motor cortex stimulation is conducted during submaximal muscle contractions (at 20% MVIC) via EMG visual feedback. Five stimuli will be delivered at each point across the grid with 5-second interval between stimuli and 1-minute rest after each point stimulation. Motor evoke potentials (MEPs) will be recorded. These MEPs will be used to represent corticospinal excitability at baseline. After completion of corticospinal excitability data collection. All electrodes will be removed, and marks on the subject's skin will be erased.

The second visit (pre-intervention visit#2) will be scheduled 1-3 day apart from the first visit (pre-intervention visit#1). Evidence demonstrates the retention of changes in cortical excitability can last for 24 hours; thus, the second visit aims to wash out the effects of TMS on corticospinal excitability from TMS measurement before receiving tDCS or NMES. LM activation measurement at baseline will be collected. The subjects will be in prone position on treatment table with thorax (T3 level) and pelvis (S2 level) securely fastened to the bed. Then, ultrasound transducer will be placed at right L4-5 facet joint by the researcher who is blinded to the group assignment. Right LM thickness at rest will be recorded. After that, the subject will be asked to perform 2 repetitions of maximum voluntary isometric contraction (MVIC) of back extension with rotation to the left to activate right LM with 1-minute rest between repetitions. The researcher will measure right LM thickness during MVIC for both repetitions. Subject will be asked to rate the rating of perceived exertion (RPE) and take 5-minute rest to prevent muscle fatigue. The neuromuscular electrical stimulation (NMES) electrodes will be placed to bilateral LM, and the system will be set at interferential mode (6000 Hz, beat frequency 20-50 Hz, scanning effect). Then, ultrasound transducer will be placed at right L4-5 facet joint by the researcher. The NMES intensity will be set at maximal tolerance to presumably activate most motor units available in the LM. The subject will be asked to perform 2 repetitions of MVIC simultaneously with the NMES.

After LM activation measurement, subjects will be randomly assigned into 3 groups (tDCS priming with MCE group, NMES priming with MCE group, and MCE alone group). For the first visit, we aim to determine the effects of tDCS and NMES against MCE. The subjects in tDCS priming with MCE group will receive the tDCS using 5X7 cm electrodes in which anodal electrode will be placed on M1 representing the back muscles (1 cm anterior and 4 cm lateral to the vertex), while cathodal electrode will be placed on contralateral supraorbital area. The intensity will be set at 2 mA with 10-second fade in/out. The subject will be stimulated by tDCS for 20 minutes. The subjects in NMES priming with MCE group will receive the NMES using interferential mode (6000 Hz, beat frequency 20-50 Hz, scanning effect) on bilateral LM. The intensity will be set at the subject's maximum tolerance. Stimulation will be set at 10 seconds on and 60 seconds off to minimize muscle fatigue. The subjects in MCE group will receive MCE for 20 minutes. After that, all subjects will undergo LM activation, lumbar stability and cortical excitability measurements using the same protocol. These data will be used to determine the immediate effects of tDCS and NMES against MCE (Objective 1 and 3). The researcher will make an appointment with the subjects for 6-week intervention program.

The 6-week intervention program can start at any day based on the subject's preference but should no longer than 1 week after baseline measurement. For 6-week intervention program, the subjects in tDCS priming with MCE group will receive a 20-minute tDCS, while the subjects in NMES priming with MCE group will receive a 20-minute NMES using the same setting as previously mentioned, and the subjects in MCE alone group will receive a 20-minute sham tDCS by setting the intensity at zero mA. After 20 minutes, the subject will receive MCE.

The subject will receive tDCS, sham-tDCS or NMES for 20 minutes followed by 20-minute supervised MCE for every session. The subject is encouraged to perform the same exercise as physical therapy session for 15 minutes once a day and keep record in the exercise logbook. The subject will receive assigned intervention twice a week for 6 weeks. The total number of interventions is 12 sessions. To increase the generalizability of the study, the researchers will not fix the day of the week. The subjects can select any days in the week that is suitable for them. However, we keep twice a week as the evidence shows improvement in pain and disability. Subjects will be asked to fill out pain and disability questionnaires, as well as undergo functional tests at week 2.

After completion of 6-week intervention program, the subjects will undergo biomechanical data collection including motion, clinical observation, LM activation, lumbar stability, and cortical excitability. Clinical outcomes including pain, disability, quality of life, fear of movement, global rating of change, as well as patient's satisfaction will be also collected. Functional tests will be performed after 6-week intervention as well. Baseline and post 6-week data will be used to compare the effectiveness of 6-week intervention program among tDCS priming with MCE, NMES priming with MCE, and MCE alone in patients with CLBP (Objective 3). In addition, corticospinal excitability, LM activation, lumbar stability, movement patterns, and clinical outcomes will be used to determine the associations among parameters (Objective 4).

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for individuals without a history of low back pain.

1. Between the ages of 18 and 40
2. No previous history of low back pain in lifetime.

The inclusion criteria for patients with CLBP individuals.

1. Between the ages of 18 and 40.
2. Having low back pain over 3 months or a recurrent pattern of LBP at least two episodes that interfered with activities of daily living and/or required treatment. This information will be obtained by interview during subjective examination.

Exclusion Criteria:

1. History of seizure for either the subject or any family member
2. Implanted pacemaker
3. Clinical signs of systemic disease
4. Definitive neurologic signs including pain, weakness or numbness in the lower extremity
5. Previous spinal surgery
6. Diagnosed osteoporosis, severe spinal stenosis, and/or inflammatory joint disease
7. Any lower extremity condition that would potentially alter trunk movement
8. Vestibular dysfunction
9. Extreme psychosocial involvement
10. Body mass index (BMI) greater than 30 kg/m2
11. Active treatment of another medical illness that would preclude participation in any aspect of the study
12. Menstruation or pregnancy (for female subject)
13. Diagnosed herniated nucleus pulposus (HNP)
14. Contraindications for TMS and tDCS including open wound, infection, lesions, arteriosclerosis, history of haemophilia or demand-type pacemaker
15. Acute cerebral hemorrhage
16. Medications that can interfere the effect of tDCS including sodium channel blocker, calcium channel blocker, NMDA receptor antagonist

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Corticospinal excitability measurement | Change from baseline after 1 session and at 6 week after intervention.
  Transcranial magnetic stimulation (TMS) will be used to measure corticospinal excitability including resting and active motor thresholds, motor evoke potentials, cortical silent period of LM, and topography (center of gravity coordinate; CoG and volume) of ES and LM, will be primary outcomes for objectives 1-4.
Muscle function measurement | Change from baseline after 1 session and at 6 week after intervention.
  Ultrasound imaging will be used to measure muscle function including TrA and LM thickness, cross-sectional area, and pennation angle will be primary outcome for objective 1-4.
Lumbar stability measurement | Change from baseline after 1 session and at 6 week after intervention.
  Electromagnetic tracking system will be used to measure spinal displacement during applying compression force to represent lumbar stability. This will be primary outcome measures for objective 1-4.
Kinematic measurement | Change from baseline at 6 week after intervention.
  Inertial measurement unit will be used to measure lumbopelvic motions during functional and clinical movement tests. These data can represent movement control. These data will be primary outcome for objectives 3 and 4.
Clinical observation of aberrant movement | Change from baseline at 6 week after intervention.
  Clinician will observe the movements and rate as presence or absence of aberrant movement.

SECONDARY OUTCOMES:
Self-report questionnaires | Change from baseline at 6 week after intervention.
  self-report questionnaires including pain, disability, quality of life, fear avoidance, global rating of change and patient's satisfaction will be secondary outcomes for objectives 3 and 4. These data will be used to describe subject characteristics and evaluate perception on provided intervention.
Functional capacity | Change from baseline at 6 week after intervention.
  Functional tests including 5-time sit to stand test (seconds), 2-minute step test (number of steps), functional reach test (centimeters), prone trunk extension test (number of repetitions) and abdominal curl test (number of repetitions) will be secondary outcomes for objectives 3 and 4.

CONTACTS AND LOCATIONS:
Overall Officials: Peemongkon Wattananon, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Physical Therapy, Mahidol University, Salaya, Changwat Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Unidentifiable data can be shared upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After December 2022 for 5 years.
Access Criteria: Written request will be reviewed by principal investigator.

REFERENCES:
- [Background] Hebert J, Koppenhaver S, Fritz J, Parent E. Clinical prediction for success of interventions for managing low back pain. Clin Sports Med. 2008 Jul;27(3):463-79, ix-x. doi: 10.1016/j.csm.2008.03.002. PMID 18503878
- [Background] Hicks GE, Fritz JM, Delitto A, McGill SM. Preliminary development of a clinical prediction rule for determining which patients with low back pain will respond to a stabilization exercise program. Arch Phys Med Rehabil. 2005 Sep;86(9):1753-62. doi: 10.1016/j.apmr.2005.03.033. PMID 16181938
- [Background] Rabin A, Shashua A, Pizem K, Dickstein R, Dar G. A clinical prediction rule to identify patients with low back pain who are likely to experience short-term success following lumbar stabilization exercises: a randomized controlled validation study. J Orthop Sports Phys Ther. 2014 Jan;44(1):6-B13. doi: 10.2519/jospt.2014.4888. Epub 2013 Nov 21. PMID 24261926
- [Background] Biely SA, Silfies SP, Smith SS, Hicks GE. Clinical observation of standing trunk movements: what do the aberrant movement patterns tell us? J Orthop Sports Phys Ther. 2014 Apr;44(4):262-72. doi: 10.2519/jospt.2014.4988. Epub 2014 Jan 22. PMID 24450372
- [Background] Laird RA, Kent P, Keating JL. Modifying patterns of movement in people with low back pain -does it help? A systematic review. BMC Musculoskelet Disord. 2012 Sep 7;13:169. doi: 10.1186/1471-2474-13-169. PMID 22958597
- [Background] Luomajoki H, Kool J, de Bruin ED, Airaksinen O. Movement control tests of the low back; evaluation of the difference between patients with low back pain and healthy controls. BMC Musculoskelet Disord. 2008 Dec 24;9:170. doi: 10.1186/1471-2474-9-170. PMID 19108735
- [Background] Hides JA, Richardson CA, Jull GA. Multifidus muscle recovery is not automatic after resolution of acute, first-episode low back pain. Spine (Phila Pa 1976). 1996 Dec 1;21(23):2763-9. doi: 10.1097/00007632-199612010-00011. PMID 8979323
- [Background] Hodges PW, Danneels L. Changes in Structure and Function of the Back Muscles in Low Back Pain: Different Time Points, Observations, and Mechanisms. J Orthop Sports Phys Ther. 2019 Jun;49(6):464-476. doi: 10.2519/jospt.2019.8827. PMID 31151377
- [Background] Kiesel KB, Underwood FB, Mattacola CG, Nitz AJ, Malone TR. A comparison of select trunk muscle thickness change between subjects with low back pain classified in the treatment-based classification system and asymptomatic controls. J Orthop Sports Phys Ther. 2007 Oct;37(10):596-607. doi: 10.2519/jospt.2007.2574. PMID 17970406
- [Background] Marshall PW, Murphy BA. Muscle activation changes after exercise rehabilitation for chronic low back pain. Arch Phys Med Rehabil. 2008 Jul;89(7):1305-13. doi: 10.1016/j.apmr.2007.11.051. PMID 18586132
- [Background] Wattananon P, Sungnak P, Songjaroen S, Kantha P, Hsu WL, Wang HK. Using neuromuscular electrical stimulation in conjunction with ultrasound imaging technique to investigate lumbar multifidus muscle activation deficit. Musculoskelet Sci Pract. 2020 Dec;50:102215. doi: 10.1016/j.msksp.2020.102215. Epub 2020 Jul 13. PMID 33220931
- [Background] Masse-Alarie H, Beaulieu LD, Preuss R, Schneider C. Influence of paravertebral muscles training on brain plasticity and postural control in chronic low back pain. Scand J Pain. 2016 Jul;12:74-83. doi: 10.1016/j.sjpain.2016.03.005. Epub 2016 May 11. PMID 28850499
- [Background] Masse-Alarie H, Beaulieu LD, Preuss R, Schneider C. Corticomotor control of lumbar multifidus muscles is impaired in chronic low back pain: concurrent evidence from ultrasound imaging and double-pulse transcranial magnetic stimulation. Exp Brain Res. 2016 Apr;234(4):1033-45. doi: 10.1007/s00221-015-4528-x. Epub 2015 Dec 26. PMID 26708518
- [Background] Silfies SP, Vendemia JMC, Beattie PF, Stewart JC, Jordon M. Changes in Brain Structure and Activation May Augment Abnormal Movement Patterns: An Emerging Challenge in Musculoskeletal Rehabilitation. Pain Med. 2017 Nov 1;18(11):2051-2054. doi: 10.1093/pm/pnx190. No abstract available. PMID 29121336
- [Background] Tsao H, Galea MP, Hodges PW. Reorganization of the motor cortex is associated with postural control deficits in recurrent low back pain. Brain. 2008 Aug;131(Pt 8):2161-71. doi: 10.1093/brain/awn154. Epub 2008 Jul 18. PMID 18669505
- [Background] Alrwaily M, Schneider M, Sowa G, Timko M, Whitney SL, Delitto A. Stabilization exercises combined with neuromuscular electrical stimulation for patients with chronic low back pain: a randomized controlled trial. Braz J Phys Ther. 2019 Nov-Dec;23(6):506-515. doi: 10.1016/j.bjpt.2018.10.003. Epub 2018 Oct 18. PMID 30482602
- [Background] Cairns MC, Foster NE, Wright C. Randomized controlled trial of specific spinal stabilization exercises and conventional physiotherapy for recurrent low back pain. Spine (Phila Pa 1976). 2006 Sep 1;31(19):E670-81. doi: 10.1097/01.brs.0000232787.71938.5d. PMID 16946640
- [Background] Ferreira ML, Ferreira PH, Latimer J, Herbert RD, Hodges PW, Jennings MD, Maher CG, Refshauge KM. Comparison of general exercise, motor control exercise and spinal manipulative therapy for chronic low back pain: A randomized trial. Pain. 2007 Sep;131(1-2):31-7. doi: 10.1016/j.pain.2006.12.008. Epub 2007 Jan 23. PMID 17250965
- [Background] Baek SO, Cho HK, Kim SY, Jones R, Cho YW, Ahn SH. Changes in deep lumbar stabilizing muscle thickness by transcutaneous neuromuscular electrical stimulation in patients with low back pain. J Back Musculoskelet Rehabil. 2017;30(1):121-127. doi: 10.3233/BMR-160723. PMID 27341642
- [Background] Hicks GE, Sions JM, Velasco TO, Manal TJ. Trunk Muscle Training Augmented With Neuromuscular Electrical Stimulation Appears to Improve Function in Older Adults With Chronic Low Back Pain: A Randomized Preliminary Trial. Clin J Pain. 2016 Oct;32(10):898-906. doi: 10.1097/AJP.0000000000000348. PMID 26736024
- [Background] Songjaroen S, Sungnak P, Piriyaprasarth P, Wang HK, Laskin JJ, Wattananon P. Combined neuromuscular electrical stimulation with motor control exercise can improve lumbar multifidus activation in individuals with recurrent low back pain. Sci Rep. 2021 Jul 20;11(1):14815. doi: 10.1038/s41598-021-94402-2. PMID 34285318
- [Background] Jafarzadeh A, Ehsani F, Yosephi MH, Zoghi M, Jaberzadeh S. Concurrent postural training and M1 anodal transcranial direct current stimulation improve postural impairment in patients with chronic low back pain. J Clin Neurosci. 2019 Oct;68:224-234. doi: 10.1016/j.jocn.2019.07.017. Epub 2019 Jul 23. PMID 31350080
- [Background] Luedtke K, Rushton A, Wright C, Jurgens T, Polzer A, Mueller G, May A. Effectiveness of transcranial direct current stimulation preceding cognitive behavioural management for chronic low back pain: sham controlled double blinded randomised controlled trial. BMJ. 2015 Apr 16;350:h1640. doi: 10.1136/bmj.h1640. PMID 25883244
- [Background] Mariano TY, Burgess FW, Bowker M, Kirschner J, Van't Wout-Frank M, Jones RN, Halladay CW, Stein M, Greenberg BD. Transcranial Direct Current Stimulation for Affective Symptoms and Functioning in Chronic Low Back Pain: A Pilot Double-Blinded, Randomized, Placebo-Controlled Trial. Pain Med. 2019 Jun 1;20(6):1166-1177. doi: 10.1093/pm/pny188. PMID 30358864
- [Background] O'Connell NE, Cossar J, Marston L, Wand BM, Bunce D, De Souza LH, Maskill DW, Sharp A, Moseley GL. Transcranial direct current stimulation of the motor cortex in the treatment of chronic nonspecific low back pain: a randomized, double-blind exploratory study. Clin J Pain. 2013 Jan;29(1):26-34. doi: 10.1097/AJP.0b013e318247ec09. PMID 23221623
- [Background] Schabrun SM, Burns E, Thapa T, Hodges P. The Response of the Primary Motor Cortex to Neuromodulation is Altered in Chronic Low Back Pain: A Preliminary Study. Pain Med. 2018 Jun 1;19(6):1227-1236. doi: 10.1093/pm/pnx168. PMID 29016867
- [Background] Schabrun SM, Jones E, Elgueta Cancino EL, Hodges PW. Targeting chronic recurrent low back pain from the top-down and the bottom-up: a combined transcranial direct current stimulation and peripheral electrical stimulation intervention. Brain Stimul. 2014 May-Jun;7(3):451-9. doi: 10.1016/j.brs.2014.01.058. Epub 2014 Jan 30. PMID 24582372
- [Background] Straudi S, Buja S, Baroni A, Pavarelli C, Pranovi G, Fregni F, Basaglia N. The effects of transcranial direct current stimulation (tDCS) combined with group exercise treatment in subjects with chronic low back pain: a pilot randomized control trial. Clin Rehabil. 2018 Oct;32(10):1348-1356. doi: 10.1177/0269215518777881. Epub 2018 May 21. PMID 29783893
- [Background] Sung W, Hicks GE, Ebaugh D, Smith SS, Stackhouse S, Wattananon P, Silfies SP. Individuals With and Without Low Back Pain Use Different Motor Control Strategies to Achieve Spinal Stiffness During the Prone Instability Test. J Orthop Sports Phys Ther. 2019 Dec;49(12):899-907. doi: 10.2519/jospt.2019.8577. Epub 2019 Aug 3. PMID 31378122
- [Background] Strutton PH, Theodorou S, Catley M, McGregor AH, Davey NJ. Corticospinal excitability in patients with chronic low back pain. J Spinal Disord Tech. 2005 Oct;18(5):420-4. doi: 10.1097/01.bsd.0000169063.84628.fe. PMID 16189454
- [Background] Tsao H, Galea MP, Hodges PW. Driving plasticity in the motor cortex in recurrent low back pain. Eur J Pain. 2010 Sep;14(8):832-9. doi: 10.1016/j.ejpain.2010.01.001. Epub 2010 Feb 23. PMID 20181504
- [Background] Agboada D, Mosayebi Samani M, Jamil A, Kuo MF, Nitsche MA. Expanding the parameter space of anodal transcranial direct current stimulation of the primary motor cortex. Sci Rep. 2019 Dec 3;9(1):18185. doi: 10.1038/s41598-019-54621-0. PMID 31796827
- [Background] O'Connell NE, Maskill DW, Cossar J, Nowicky AV. Mapping the cortical representation of the lumbar paravertebral muscles. Clin Neurophysiol. 2007 Nov;118(11):2451-5. doi: 10.1016/j.clinph.2007.08.006. Epub 2007 Sep 24. PMID 17890149
- [Background] Tsao H, Danneels LA, Hodges PW. ISSLS prize winner: Smudging the motor brain in young adults with recurrent low back pain. Spine (Phila Pa 1976). 2011 Oct 1;36(21):1721-7. doi: 10.1097/BRS.0b013e31821c4267. PMID 21508892